CLINICAL TRIAL: NCT07174297
Title: To Compare the Efficacy and Safety of Acotiamide Versus Itopride in Patient With Post Prandial Distress Syndrome Type of Functional Dyspepsia
Brief Title: Acotiamide vs Itopride in Postprandial Distress Syndrome
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Collaborators: Rawalpindi Medical College, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GTZ-FD-012-25
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postprandial Distress Syndrome
MeSH Terms: interventions — Z 338; itopride

STUDY DESIGN:
Intervention Model Description: Open-label, comparative randomized, parallel, two-arms, multi-center study. A permuted block randomization technique was applied to generate an individual list of random assignment of participants to treatment group A (Acotiamide) and treatment group B (Itopride). A block represents a separate center/site of enrollment, and each center will enroll total 50 - 55 participants as per protocol. There will be total 3 recruitment centers, and each recruiting center will follow the provided list of random assignments (Annexure). An online software (https://www.sealedenvelope.com/simple-randomiser/v1/lists) was used to generate a random sequence for total 152 subjects with balanced distribution method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- assignment of participants to treatment group A (Acotiamide) (Active Comparator)
  Interventions: Drug: Acotiamide
- assignment of participants to treatment group B (Itopride). (Active Comparator)
  Interventions: Drug: Acotiamide

INTERVENTIONS:
Drug: Acotiamide — Both these drugs are used for the management of PDS type of FD
  Other Names: Itopride

SUMMARY:
The goal of this study is to "To compare the efficacy and safety of Acotiamide versus Itopride in patient with post prandial distress syndrome type of functional dyspepsia"

DETAILED DESCRIPTION:
Investigator is aiming to conduct an Open-label, comparative randomized controlled, parallel, two-arms, multi-center study.

Primary Outcomes:

• Difference in overall treatment effect between both groups by using Leuven Postprandial Distress Scale (LPDS) in 8 weeks from the baseline

Secondary Outcomes:

* Difference between both groups in symptoms of Postprandial Distress Syndrome (PDS) (including early satiety, abdominal bloating, postprandial fullness) by using Leuven Postprandial Distress Scale (LPDS)
* Difference between both groups in quality of life by using short form Nepean Dyspepsia Index (SF-NDI) from baseline
* Frequency of adverse events, serious adverse events and tolerability in both groups

ELIGIBILITY:
Inclusion Criteria:

* Subjects to provide written informed consent prior to any study procedures being performed
* Subjects with age 18-70 both male and female
* Diagnosed with FD (PDS) by using ROME IV criteria
* Subjects naive to acotiamide and Itopride for last 2 weeks
* Subjects must have a normal endoscopy result within the 6 months

Exclusion Criteria:

* Without predominant symptoms of ulcer and GERD based on history & endoscopy, IBS based on history & Rome IV criteria and Chronic idiopathic nausea based on history only
* Subjects taking drugs that affect gut motility, gut sensitivity, SSRI and/or acid secretion who are unable to discontinue these drugs before initiating the intervention
* Subjects with chronic medical disorders potentially contributing to PDS such as chronic pancreatitis, hypothyroidism, CKD and CLD identified through clinical history, physical examination, or previous medical records
* Subjects with Type I or Type II diabetes
* Pregnant & lactating mothers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference in overall treatment effect between both groups by using Leuven Postprandial Distress Scale in 8 weeks | 8 weeks
  Overall treatment effect will be assessed using the Leeds Postprandial Distress Scale, with change in total score from baseline before initiation of treatment end of treatment. The decreased score representing the treatment response.

SECONDARY OUTCOMES:
Difference between both groups in symptoms of Postprandial Distress Syndrome (PDS) (including early satiety, abdominal bloating, postprandial fullness) by using Leuven Postprandial Distress Scale | 8 weeks
  All the symptoms of PDDS will be assessed by using the Leeds Postprandial Distress Scale (LPDS), with change in total score from baseline before treatment initiation to end of treatment going downwards representing the treatment response.
Difference between both groups in quality of life by using short form Nepean Dyspepsia Index scale | 8 weeks
  Quality of life will be assessed using the Nepean Dyspepsia Index, defined as the change in total score from baseline to the end of the treatment with lower scores indicating improvement
Frequency of adverse events, serious adverse events and tolerability in both groups | 8 weeks
  Frequency of adverse events will be assessed through a patient diary maintained throughout the study, with entries reviewed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muahmmad Umar, MBBS, FCPS, FACG, AGAF, FRCP, Principal Investigator — Rawalpindi Medical University/College

IPD SHARING:
Plan to Share IPD: Undecided
it will be decided after closing of enrollment